CLINICAL TRIAL: NCT03545464
Title: COrticosteroids in acUte uRticAria in emerGency dEpartment
Acronym: COURAGE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P160913J
Record Dates: First submitted 2018-04-13; First posted 2018-06-04 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Urticaria; Angiœdema
Keywords: Acute urticaria
MeSH Terms: conditions — Urticaria | interventions — Prednisone; levocetirizine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Antihistamines + placebo of cortancyl (Experimental): - In emergency department : Levocetirizine 5 mg orally. Renewable once if persistence of hives at 30 minutes.
  Placebo of Cortancyl : 1mg/kg (the number of tablets the patient needs to take is based on his weight and is noted on annex 4), once orally
  - At home : Levocetirizine 5 mg twice daily for 7 days (D1 to D7). If persistence of hives, levocetirizine 10 mg twice daily for 7 more days (D8 to D14).
  Placebo of Cortancyl 20 mg x 2 tablets = 40mg once per day for 3 days orally
  Interventions: Drug: Placebo Oral Tablet; Drug: Levocetirizine Oral Tablet
- Association of antihistamines and cortancyl (Active Comparator): - In emergency department : Levocetirizine 5 mg orally Renewable once if persistence of hives at 30 minutes.
  Cortancyl: 1 mg/kg (the number of tablets the patient needs to take is based on his weight and is noted on annex 4), once orally.
  - At home : Levocetirizine 5 mg twice daily for 7 days (D1 to D7). If persistence of hives, levocetirizine 10 mg twice daily for 7 more days (D8 to D14).
  Cortancyl : 20 mg x 2 tablets = 40 mg per day for 3 days orally
  Interventions: Drug: Cortancyl Oral Tablet; Drug: Levocetirizine Oral Tablet

INTERVENTIONS:
Drug: Placebo Oral Tablet — Placebo of cortancyl Oral Tablet 20mg
  Arms: Antihistamines + placebo of cortancyl
Drug: Cortancyl Oral Tablet — Cortancyl oral Tablet 20 mg
  Arms: Association of antihistamines and cortancyl
Drug: Levocetirizine Oral Tablet — Levocetirizine Oral Tablet 5 mg

SUMMARY:
To demonstrate the non-inferiority of the efficacy of a single antihistamine in comparison with an association of antihistamine and corticosteroid in the treatment of acute urticaria in emergency departments

DETAILED DESCRIPTION:
Acute urticaria (hives) is a common skin disease. The prevalence of acute urticaria in life is about 15 to 20% in the general population. It is responsible for a frequent use of emergency departments (ED). The usual treatment is based on early administration of an association of antihistamines and corticosteroid. The therapeutic efficacy of corticosteroids has never been established by high evidence studies. However, corticosteroids are frequently used. When stopped, corticosteroids could promote the occurence of urticaria recurrences, and a transition to chronic urticaria. In addition, corticosteroids may be rarely responsible for gastrointestinal bleeding, hypertension and diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Isolated acute urticaria (acute hives): spontaneous urticaria, inducible urticaria
* Acute urticaria with angioedema without laryngeal edema
* Obtain patient's consent
* Social security affiliation

Exclusion Criteria:

* Pregnancy or breastfeeding
* Acute hives with anaphylaxis
* Bradykinin angioedema
* Angioedema without urticaria (hives)
* Laryngeal edema with urticaria (hives)
* Corticosteroid administration in the previous 5 days visiting the emergency department
* Antihistamines greater than 1 tablet per day in the previous 5 days visiting the ED
* Other treatment for urticaria : omalizumab, montelukast, ciclosporin A
* Chronic urticaria before acute urticaria diagnosis
* Atopic dermatitis
* Eczema
* Bullous pemphigoid
* Acute exanthematous pustulosis
* Diabetes mellitus
* Gastrointestinal ulcer
* Refusal to participate
* Known allergy to the study drugs or formulation ingredients
* Known Renal failure defined by creatinine clearance < 10 mL/min or cardiac failure defined by ejection fraction < 40%.
* Corticoid use in 5 days prior to randomisation
* Contra-indication to corticotherapy:
* Any live vaccine
* Psychotic states still uncontrolled by treatment limiting the participant's compliance with the research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 137 (Actual)
Dates: Start 2019-09-21 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-09-17 (Actual)

PRIMARY OUTCOMES:
7-Days Urticaria Activity Score (UAS 7) at day 7 | For 7 day
  Urticaria Activity Score (UAS) is a daily combined score of severity of itch and number of hives. Each component of the UAS is scored on a scale of 0 to 3; the 2 scores are added together for a daily total of 0 to 6.

SECONDARY OUTCOMES:
Recurrence of hives at day 7 and/or recurrence of itch at day 7 | For 7 day
  The UAS 7 is the sum of the daily UAS scores over 7 days. This questionnaire will be completed by the patient and the investigator.
Occurrence of spontaneous wheals and/or itch for > 6 weeks | beyond 6 Weeks
  wheals and/or itch for > 6 weeks
Patients with angioedema at day 7, 14 and 3 months | up to 3 month
  angioedema
The reduction of morbidity is assessed by new emergency visits for acute urticaria recurrences at day 7, 14 and 3 months | up to 3 month
  emergency visits
(DLQI) up to 6 months | up to 6 months
  The DLQI is a dermatology-specific quality of life questionnaire designed for use in patients over 16 years of age
Cu-Q2QoL up to 6 months | at day 7, at day 14, at 6 week, at 3 months and 6 months
  The CU-Q2oL (French version) is a questionnaire that measures the relative burden of chronic urticaria on subjective well-being

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas JAVAUD, M.D,Ph.D, Principal Investigator — France Hospital Louis MOURIER Colombes, Ile De France, France, 92700
Locations (1):
- Hospital Louis MOURIER, Colombes, Île-de-France Region, France

REFERENCES:
- [Derived] Javaud N, Soria A, Maignan M, Martin L, Descamps V, Fain O, Bouillet L, Berard F, Tazarourte K, Roy PM, Fontaine JP, Bagot M, Khellaf M, Goulet H, Lapostolle F, Casalino E, Doutre MS, Gil-Jardine C, Caux F, Chosidow O, Pateron D, Vicaut E, Adnet F. Glucocorticoids for acute urticaria: study protocol for a double-blind non-inferiority randomised controlled trial. BMJ Open. 2019 Aug 21;9(8):e027431. doi: 10.1136/bmjopen-2018-027431. PMID 31439599